CLINICAL TRIAL: NCT06160804
Title: Evaluating Skeletal Traction for Patients With Femoral Shaft Fractures Treated With Intramedullary Nailing Within 24 Hours of Presentation
Brief Title: Evaluating Femoral Traction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolling subjects intro the trial was difficult. It would not have been possible to complete the study within a reasonable timeline based on the current enrollment.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0183
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-05

CONDITIONS: Femoral Shaft Fracture

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Subgroups will be determined using equal block randomization. Block randomization will be used for this study. Blocks will be set to groups of 4 with each block of 4 comprising 2 traction and 2 splint opaque envelopes in random order. The envelope will be stored in the office of the principle investigator and opened following subject enrollment. This ensures subjects are blinded to their initial treatment modality. Standard of care will be followed for all clinical decisions beyond the type of stabilization procedure to be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local standard of care (Placebo Comparator)
  Interventions: Procedure: Skeletal traction
- Experimental change in care (Active Comparator)
  Interventions: Procedure: Femoral shaft splinting

INTERVENTIONS:
Procedure: Skeletal traction — A pin through the bone with weights attached
  Arms: Local standard of care
Procedure: Femoral shaft splinting — A splint of the broken thigh bone
  Arms: Experimental change in care

SUMMARY:
The primary goal of this study is to test the hypothesis that skeletal traction allows for easier intraoperative reduction time by comparing the reduction time in patients that receive skeletal traction for femoral shaft fracture to those that do not. Secondary goals are to assess the claims of improved pain control and decreased blood loss in patients that receive skeletal traction for femoral shaft fracture to those that do not.

DETAILED DESCRIPTION:
Traction is a practice dating back thousands of years, historically used for the definitive treatment of femoral shaft fractures. With advances in surgical care, traction is no longer regularly used for definitive treatment. However, traction is commonly used preoperatively with the claimed benefits of fracture stabilization allowing for improved pain control, restoration of limb length with easier operative reduction, and controlling bleeding by decreasing compartmental volume. However, studies have begun to question the utility of skeletal traction in patients with femoral shaft fractures.

While pre-hospital traction splints may provide added pain control for patients with femoral shaft fractures as they are transported to the hospital, skeletal traction may not provide the same pain control benefits in the inpatient setting. Dr. Bumpass and colleagues prospectively compared patients with femoral shaft fractures placed into distal femoral traction to those that were splinted. The authors demonstrated that while patients that were splinted reported higher pain scores during application, pain scores after immobilization were not different between the two groups.

Retrospective and prospective investigations of traction for femoral shaft fractures have failed to demonstrate easier operative reduction or decreased blood loss. Koerner et al retrospectively evaluated patients with femoral shaft fractures that underwent definitive intramedullary nailing within 24 hours of presentation. The authors demonstrated no difference in blood loss, transfusion requirement, or need for open reduction between patients placed in skeletal traction and patients placed in lower extremity splints. Similarly, in their randomized controlled trial Even et al demonstrated no difference in reduction time for patients with femoral shaft fractures fixed within 24 hours that received skeletal traction or skin traction preoperatively.

To the investigator's knowledge, no study has prospectively compared surgical time, pain control, and blood loss for patients that receive preoperative skeletal traction to splinting for femoral shaft fractures that receive intramedullary nailing within 24 hours of presentation.

Skeletal traction has a long history in orthopaedic surgery for the treatment of femoral shaft fractures, but may be unnecessary for patients that are surgically treated within 24 hours of presentation. The primary goal of this study is to test the hypothesis that skeletal traction allows for easier intraoperative reduction time by comparing the reduction time in patients that receive skeletal traction for femoral shaft fracture to those that do not. Secondary goals are to assess the claims of improved pain control and decreased blood loss in patients that receive skeletal traction for femoral shaft fracture to those that do not.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient (ages 18 and over) with a femoral shaft fracture that is treated with intramedullary nailing within 24 hours of presentation

Exclusion Criteria:

* Patients younger than 18
* Polytraumatized patients
* Patients with pathological fractures
* Patients with femoral shaft fracture not amenable to intramedullary nailing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Time to reduce a femoral shaft fracture | Within 24 hours of presentation
  Time to reduce a femoral shaft fracture is decreased in patients that receive preoperative traction. Time measured in minutes. Short time means faster time to reduction.

SECONDARY OUTCOMES:
Change in preoperative opiate requirement | 24 hours from presentation
  To see if Patients that receive preoperative traction for a femoral shaft fracture have a change in preoperative opiate requirement as measured by morphine equivalents/kg/hr. More morphine means lower pain control.
Change in transfusion requirement | Within 24 hours of presentation
  To determine if patients that receive preoperative traction for a femoral shaft fracture have a change in transfusion requirement. Measured by total liters of blood given to patient during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Christiano, MD, Principal Investigator — University of Chicago faculty
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared

REFERENCES:
- [Background] Obey MR, Berkes MB, McAndrew CM, Miller AN. Lower-Extremity Skeletal Traction Following Orthopaedic Trauma: Indications, Techniques, and Evidence. JBJS Rev. 2019 Nov;7(11):e4. doi: 10.2106/JBJS.RVW.19.00032. No abstract available. PMID 31764196
- [Background] Even JL, Richards JE, Crosby CG, Kregor PJ, Mitchell EJ, Jahangir AA, Tressler MA, Obremskey WT. Preoperative skeletal versus cutaneous traction for femoral shaft fractures treated within 24 hours. J Orthop Trauma. 2012 Oct;26(10):e177-82. doi: 10.1097/BOT.0b013e31823a8dae. PMID 22430522